CLINICAL TRIAL: NCT00702429
Title: Immunoregulation of Periodontal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2007-A00632-51
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Periodontal Disease
MeSH Terms: conditions — Periodontal Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients achieve of parodontopathies
  Interventions: Other: Blood sampling
- 2 (Placebo Comparator): Patients without parodontales diseases
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Analysis of the PNN, analysis of the monocytes
  Arms: 1
Other: Blood sampling — Analysis of the PNN, analysis of the monocytes
  Arms: 2

SUMMARY:
Our design is to test in hospital practice a selection of immune parameters that could assess the pathophysiology and progression of periodontal lesions.

DETAILED DESCRIPTION:
These parameters will be measured in 25 healthy volunteers and 25 moderate-to severe periodontal disese patients. Phagocytes will be tested phenotypically and functionally, both ex vivo and in vitro.

ELIGIBILITY:
Inclusion Criteria:

* Persons appearing spontaneously at the consultation of parodontologie for parodontale disease,
* persons agreeing to undergo a sampling of blood intended for the search

Exclusion Criteria:

* Presence of a chronic or pointed pathology,
* an age 18-year-old subordinate or 65-year-old superior,
* pregnant women,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Percentage of positive cells and intensity of expression for the molecules of surface studied there cytometric in stream | 24 months

SECONDARY OUTCOMES:
Rate of secretion of cytokines and the other substances | 24 months
Detection and quantification of ARN messengers | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Joana VITTE, MD, Principal Investigator — Assistance Publique des Hôpitaux de Marseille
Locations (1):
- Hopital de la Conception- Laboratoire d'Immunologie, Marseille, France